CLINICAL TRIAL: NCT00500877
Title: Mood Management Phone Counseling in Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA017947 (NIH); R01DA017947 (NIH)
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Cigarette Smoking
Keywords: Smoking cessation; Phone Counseling
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mood Management Phone counseling (Active Comparator): Mood management phone counseling for smoking cessation
  Interventions: Behavioral: Mood Management Phone Counseling for Smoking Cessation
- Phone Counseling Standard (Placebo Comparator): Phone counseling standard
  Interventions: Behavioral: Mood Management Phone Counseling for Smoking Cessation

INTERVENTIONS:
Behavioral: Mood Management Phone Counseling for Smoking Cessation — Phone counseling addressed mood management and smoking cessation

SUMMARY:
Information obtained from this study will help us to have a better idea of how phone counseling may facilitate the process of quitting smoking for individuals with a history of recurrent depression.

DETAILED DESCRIPTION:
Adult smokers with a history of recurrent major depression (MDD) report higher levels of depressive symptoms when presenting for smoking cessation treatment and have poor smoking outcomes relative to other smokers. Carefully conducted clinical trials have supported the efficacy of cognitive-behavioral mood management treatment for depression in improving smoking cessation outcomes in this high-risk group. Although efficacious, these intensive group treatments require significant resources and thus may have limited impact outside of specialized smoking cessation programs. In the present study we will develop and obtain preliminary data on the efficacy of proactive telephone counseling for smoking cessation that integrates cognitive-behavioral mood management skills training for depression (MM). Smokers with a history of recurrent MDD will be randomly assigned to the proactive telephone counseling for smoking cessation with mood management (MM) or a standard proactive telephone counseling (ST) comparison condition. We expect that this program of research will result in the development of a specialized, efficacious treatment with broad reach into a significant subpopulation of smokers at greatest risk for difficulties quitting, and will therefore have important clinical and public health significance in decreasing the overall prevalence of cigarette smoking.

ELIGIBILITY:
Inclusion Criteria:

* history of two or more past episodes of depression
* regular cigarette smoker for at least one year
* currently smoking 10 or more cigarettes each day
* want to quit smoking

Exclusion Criteria:

* Current Depressive Episode
* Current Alcohol of Substance abuse
* Pregnant, planning to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Smoking Abstinence | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Strong, Ph.D., Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States